CLINICAL TRIAL: NCT01934270
Title: Growth Hormone Secretion Following the Anaerobic Exercise
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Dan Nemet, MD, Prof. of Pediatric, MD, Meir Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MeirMc094-13CTIL
Record Dates: First submitted 2013-08-19; First posted 2013-09-04 (Estimated); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Short Stature; Obesity, Childhood
MeSH Terms: conditions — Dwarfism; Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Anaerobic Test (Experimental)
  Interventions: Other: Anaerobic Test

INTERVENTIONS:
Other: Anaerobic Test — To evaluate the secretion of growth hormone in response to anaerobic exercise in children.

SUMMARY:
Proper growth in children is a complex process regulated by a combination of genetic, nutritional, environmental, hormonal, and others. Growth hormone (GH) is the main hormone regulating the growth from childhood to adulthood. Despite great progress in the field, with the development of recombinant GH for the treatment of growth hormone deficiency (GHD), there is still no reliable method for testing GHD. Physical exertion is one of the significant physiologic stimuli for GH secretion, and it is reliable test for identification of GHD. It is not in use in the clinics because of its complexity. Recently GH secretion following short anaerobic exercise in young adults was tested and also demonstrated significant growth hormone secretion

In contrast to adult children's exercise is characterized by an anaerobic nature. There is no data about secretion of growth hormone in response to anaerobic exercise in children.

Purpose of the experiment:

The purpose of this study is to evaluate the secretion of growth hormone in response to anaerobic exercise in children.

DETAILED DESCRIPTION:
100 children aged 6-16 years, followed at the pediatric endocrinology clinic for growth assessment or obesity. Assessment of their growth hormone axis will be evaluate in parallel according to the currently accepted pharmacological GH testing as accepted and also following anaerobic physical test.

After explanation to the patient and his parent and obtaining an informed consent, the children will be instructed to pedal at maximum speed for 15 seconds x 10 sprints (1 minute of recovery between the sprints) against a resistance adjusted according to their body mass index.

The test will perform in similarity to GH provocative protocols by mean that they will be performed in the morning after a night's sleep and overnight fasting. The patients will be remained fasting during the test.

They will be asked not to exercise a day before the test. Thirty minutes before the test, Venflon will be inserted and the child will receive an explanation and rest until the beginning of the test. blood GH, IGF-1, cortisol will be taken at the beginning of exercise (time 0), at the end of exercise, after 30 minutes, 45 minutes and 60 minutes is customary according to criteria set pharmacological inventory growth hormone.

The test results will be compared to pharmacological testing of the child if available.

ELIGIBILITY:
Inclusion Criteria:

* Children evaluated for short stature
* Normal weight \ overweight \ obesity

Exclusion Criteria:

* Known GH deficiency

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2014-05 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Growth Hormone Release | GH will be measured at the beginning of exercise (time 0), and the change in GH level will be assessed at the end of exercise (30 seconds), after 10 minutes, 30 minutes and 60 minutes

SECONDARY OUTCOMES:
IGF-1 and Cortisol Release | IGF-1, Cortisol will be taken at the beginning of exercise (time 0), at the end of exercise (30 seconds), after 10 minutes, 30 minutes and 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Dan Nemet, MD, Principal Investigator — Meir Medical Center , Tel Aviv University
Locations (1):
- Meir Medical Center, Kfar Saba, Israel